CLINICAL TRIAL: NCT05982119
Title: Gait Analysis Parameter, Stair Climbing and Upper Limb Evaluation in Patients With Muscular Pathology and in Control Subjects: The ActiLiège Next Study
Brief Title: Assessments in Patients With Muscular Pathology and in Control Subjects : The ActiLiège Next Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Collaborators: SYSNAV (Industry)
Responsible Party: Principal Investigator, Laurent Servais, Professor Laurent Servais, Centre Hospitalier Universitaire de Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ActiLiege Next
Record Dates: First submitted 2021-07-20; First posted 2023-08-08 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Duchenne Muscular Dystrophy; Fascioscapulohumeral Muscular Dystrophy; Myotonic Dystrophy 1; Charcot-Marie-Tooth; Centronuclear Myopathy; Congenital Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophy, Facioscapulohumeral; Myotonic Dystrophy; Charcot-Marie-Tooth Disease; Myopathies, Structural, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with DMD/FSHD/CMT/DM1/CNM/FKRPmutation or control subjects (Other): Patients and control subjects will be included over a 3-years study period. Patients will be examined by a neuropaediatrician or neurologist and perform standardized assessments (timed tests, motor function tests, and strength tests) at baseline and then every 6 to 12 months (depending on age).
  From February 2024, controls subjects can be remotely recruited and enrolled. They won't be evaluated on site, but data, such as age, sex, weight, and height, will be collected by phone or visio-conference at inclusion and every 6 months for 3 years.
  Patients will be asked to wear the device during 1 to 3 months at baseline (depending on disease group) and then for 1 month every 3-12months (depending on age and disease group).
  Control subjects will be examined by a physician and perform the same tests than those for ambulant patients at baseline and 12 months. Control subjects will be asked to wear the device for two months (one month at inclusion, one month 11 months after inclusion).
  Interventions: Device: ActiMyo/Syde

INTERVENTIONS:
Device: ActiMyo/Syde — The two "watches" can be worn as wristwatch or placed near the ankle and on the wheelchair.
  * Patients with DMD or FKRP mutation will wear the ActiMyo°/Syde° during 3 months at baseline and then for one month every 3 months.
  * Patient with FSHD, DM1, CMT, CNM will wear the ActiMyo°/Syde° will wear the ActiMyo/Syde° during 3 months at baseline and then for one month every 6 months.
  * Control subjects >4years will wear the ActiMyo°/Syde° during one month after inclusion and during one other month 11 months after inclusion.
  * Control subjects <4years will wear the ActiMyo°/Syde° during one month after inclusion and during one other month every 6months after inclusion.

SUMMARY:
The objective of the ActiLiège Next study is to collect longitudinal data from patients and control subjects using a wearable magneto-inertial device. By collecting natural history data in various neuromuscular disorders (Duchenne Muscular Dystrophy, Fascioscapulohumeral Muscular Dystrophy, Myotonic Dystrophy 1, Charcot-Marie-Tooth, Centronuclear Myopathy, Congenital Muscular Dystrophy), we aim to validate digital outcome measures to continuously assess motor function in real-life.

ELIGIBILITY:
Inclusion criteria

* For the patients:

  * Genetically confirmed diagnosis of DMD, FSHD, DM1, CMT or FKRP mutations or confirmed CNM based on muscle biopsy.
  * FSHD, DM1, CMT and CNM patients should be ambulant or in transition.
  * DM1 and CMT patients should present sensori-motor signs on physical examination.
  * Under the age of 20 years for patients with DMD, CNM or between the ages of 5 and 80 years for patients with FSHD, CMT and DM1.
  * More than 2 years old for patients with FKRP mutations
  * Non-ambulant DMD patients must be able to remain seated in an arm- or a wheelchair for at least one hour.
  * Patients with DMD treated with corticosteroids for at least 6 months or initiated corticosteroid at V0 (except for patients under 4).
  * Signed informed consent form by patient himself or, in case of minor patients, signed informed consent form by patient's parents or legal guardians.
* For the control subjects:

  * Ambulant boys and girls under 20 years old
  * Signed informed consent form by patient him/herself or, in case of minor patients, signed informed consent form by patient's parents or legal guardians.

Exclusion Criteria:

* For the patients:

  * Patients with extreme cognitive disorders that limit their understanding of the exercises to be performed.
  * Patients who have undergone a surgical procedure or who have experienced recent trauma (within fewer than 6 months) affecting the upper or lower limbs (for ambulant patients).
  * A concomitant chronic or acute neurological, endocrine, infectious, allergic, or inflammatory pathology within the 3-week period immediately prior to inclusion.
  * Patients who are participating in an interventional clinical trial.
  * DMD patients in transition who are not on corticosteroids.
* For the control subjects:

  * Patients who have undergone a surgical procedure or who have experienced recent trauma (within fewer than 6 months) affecting the upper or lower limbs.
  * Elite athletes (at the national level).
  * A chronic or acute muscular, neurological, infectious, or inflammatory pathology within the 3-week period immediately prior to inclusion.
  * An orthopedic, neuromuscular, or neurological pathology that affects the quality of the subject's walking gait.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Stride velocity | through study completion (3 year)
  Stride velocity obtained with a magneto-inertial sensor (Actimyo°) in real-life (meter per second).
Stride length | through study completion (3 year)
  Stride length obtained with a magneto-inertial sensor (Actimyo°) in real-life (meter).
Stairs number | through study completion (3 year)
  Total number of strides in stairs obtained with a magneto-inertial sensor (Actimyo°) in real-life
Stairs speed | through study completion (3 year)
  Vertical speed during strides in stairs obtained with a magneto-inertial sensor (Actimyo°) in real-life
Stairs height | through study completion (3 year)
  Height of the strides in stairs obtained with a magneto-inertial sensor (Actimyo°) in real-life

CONTACTS AND LOCATIONS:
Locations (8):
- CHR de la Citadelle, Liège, Belgium
- Fakultni nemocnice v Motole, Prague, Czechia
- Galaa Military Medical Complex, Cairo, Egypt
- Semmelweis University 2nd Department of Paediatrics, Budapest, Hungary
- Warsaw Medical University Hospital, Department of Neurology, Warsaw, Poland
- Romania (2):
  - Pediatric Neurology Clinic, Clinical Hospital of Psychiatry "Prof. Dr. Al. Obregia", Bucharest
  - National Clinical Hospital for Children Neurohabilitation "Dr Nicolae Robanescu", Bucharest
- University Children's Hospital, Department for Pediatric Neurology, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No